CLINICAL TRIAL: NCT01382056
Title: Effects of Pulse Varieties on Blood Vessel Function in Individuals With Peripheral Artery Disease (PAD)
Brief Title: Effects of Pulse Varieties on Blood Vessel Function in Peripheral Artery Disease
Acronym: PULV-2011
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Pulse Canada (Other)
Responsible Party: Principal Investigator, Dr. Peter Zahradka, Professor, Department of Physiology, University of Manitoba
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: B2011:026
Record Dates: First submitted 2011-06-22; First posted 2011-06-27 (Estimated); Last update posted 2014-02-12 (Estimated); Status verified 2014-02

CONDITIONS: Peripheral Artery Disease
Keywords: Peripheral Artery Disease; Pulses; Beans; PAD
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Mixed beans (higher amount) (Experimental): Participants may be randomized to foods containing 0.6 cup of mixed beans daily 5 times per week for 8 weeks
  Interventions: Other: Mixed bean (higher amount)
- Mixed beans (lower aomunt) (Experimental): Participants may be randomized to foods containing 0.3 cup of mixed beans daily, 5 times per week for 8 weeks.
  Interventions: Other: Mixed beans (lower amount)
- Control foods (Active Comparator): pulse-free control foods consumed daily, 5 days per week for 8 weeks
  Interventions: Other: control foods

INTERVENTIONS:
Other: control foods — pulse-free control foods consumed daily, 5 days per week for 8 weeks
  Arms: Control foods
Other: Mixed bean (higher amount) — 0.6 cup of mixed beans consumed 5 days per week for 8 weeks
  Arms: Mixed beans (higher amount)
Other: Mixed beans (lower amount) — 0.3 cup of mixed beans consumed daily, 5 days per week for 5 weeks
  Arms: Mixed beans (lower aomunt)

SUMMARY:
Consumption of a diet containing pulse crops provides flavonoid compounds that will improve vascular function and glycemic control in individuals with Peripheral Artery Disease.

DETAILED DESCRIPTION:
This is a single site, randomized, controlled, food intervention study designed to explore the effects of pulse types and varieties on blood vessel function in individuals with Peripheral Artery Disease.

Phase One(Acute): To identify relative potency of pulse types (beans,peas, lentils,and chickpeas) for vascular activity in healthy participants and participants with Peripheral Artery Disease. Healthy participants (10) and participants with Peripheral Artery Disease (10) will be asked to consume (in random order) one test food per in-person visit over 5 visits scheduled a minimum of 6 days apart. Vascular responsiveness will be monitored non-invasively by peripheral arterial tonometry before consumption of the test food and 2 hours post food consumption. Blood samples will be collected at the same time intervals for analyses, of vascular, inflammatory, and metabolic markers as well as flavonoids present in the pulses.

Phase Two(Chronic): Chronic 8-week study using mixed beans (pinto, kidney, black, and navy) to determine improvements in vascular function, cardiovascular risk factors, and glycemic control in participants with Peripheral Artery Disease (N=75, 25/group). Participants will be randomly assigned to one of the following three groups: i) foods containing 0.6 cup mixed beans/day consumed 5 days per week (total amount is 3 cups mixed beans per week); or, ii) foods containing 0.3 cup mixed beans/day for 5 days per week); or, iii) pulse-free foods (control) consumed 5 days/week. A total of 3 in-person visits for screening, baseline and final will be required during the 8-week study schedule. Assessments of vascular function, cognitive function, food dietary intake and preferences, flavonoid levels and cardiovascular risk markers in blood and urine, glycemic control, and anthropometrics will be completed at baseline and at 8 weeks.

Phase Three(Follow-Up: An 8-week follow-up assessment with a subset of participants (n=10/group, 3 groups) with Peripheral Artery Disease will be done at 2, 4, and at 8 weeks. Assessments of vascular function, cognitive function, food dietary intake, flavonoid levels and cardiovascular risk markers in blood and urine, glycemic control, and anthropometrics will be completed. These assessments will enable us to determine the length of time the benefits of the pulse consumption are retained.

ELIGIBILITY:
Inclusion Criteria:

Healthy Participants, Acute Phase:

* Healthy volunteers, male or female, >33 years of age, age matched with PAD participants ± 7 years;
* BMI 18-30;
* Glycated hemoglobin < 6.5%;
* Fasting serum total cholesterol < 4 mmol/L and triglycerides < 2.5 mmol/L;
* Blood pressure < 140/90 mm Hg;
* Ankle-brachial Index (ABI) >0.9;
* Willing to comply with the protocol requirements;
* Willing to provide informed consent.

Inclusion Criteria, Participants with Peripheral Artery Disease (Acute Phase and Chronic Phase):

* Male or female, > 40 years of age;
* Documented Peripheral Artery Disease including those with claudication as defined by an ankle brachial Index of ≤ 0.90; or asymptomatic carotid stenosis of > 50% or confirmed by imaging; or having had a previous intervention for Peripheral Artery Disease or carotid disease;
* Stable medication profile with no changes required for the past 3 months;
* Willing to comply with the protocol requirements;
* Willing to provide informed consent.

Exclusion Criteria:

Healthy Participants, Acute Phase:

* Currently smoking, or smoking within the last 6 months;
* Clinically diagnosed disease affecting the heart, liver, kidneys, lungs, gastrointestinal, endocrine or blood/immune systems that requires medical treatment;
* Taking any prescribed medication with the exception of birth control and hormone (estrogen) replacement therapy;
* Pregnancy;
* Amputation of upper or lower extremity on both sides;
* History of severe gastrointestinal reactions or allergies to pulses or ingredients used to prepare the pulse-containing and pulse-free foods.

Exclusion Criteria, Participants with Peripheral Artery Disease (Acute Phase and Chronic Phase):

* Currently smoking, or smoking within the last 6 months;
* Type 1 diabetes;
* Renal failure requiring dialysis;
* Acute cardiovascular event or medical illness within the past 3 months precluding study participation;
* Hormone (estrogen) replacement therapy;
* Amputation of upper or lower extremity on both sides;
* History of severe gastrointestinal reactions or allergies to pulses or ingredients used to prepare the pulse-containing and pulse-free foods;
* Currently participating in or having participated in a food study within the last 3 months unless randomized to a control group and consumed no study foods;
* High pulse consumption (greater or equal to 2 servings per week);
* Inability to adhere to a regular diet;
* Additional intake of pulses other than the requirements outlined in the study.

Min Age: 34 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2012-03; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Evaluate individual pulse types and varieties in healthy participants and participants with Peripheral Artery Disease. | 5-week schedule
  Vascular responsiveness will be monitored non-invasively by peripheral arterial tonometry before consumption of the test food and 2 hours post food consumption. Blood samples will be collected at the same time intervals for analyses, of vascular, inflammatory, and metabolic markers as well as flavonoids present in the pulses.

SECONDARY OUTCOMES:
Evaluate the effects of mixed beans to determine improvements in vascular function | 16 weeks
  Ankle brachial index, blood vessel function and claudication onset/walking distance will be measured and compared at the pre/post consumption time points (time 0, Week 8) in participants receiving food items with the most potent pulse variety or the control food items, and in follow-up during the post consumption follow-up phase at Weeks 2,4, and 8. Results of blood samples will be assessed and compared at the same time points for lipids, glucose, insulin, glycated hemoglobin and select markers of vascular function.
Analysis of dietary patterns and nutritional intake, compliance and tolerability before and after consumption of an 8-week diet of mixed beans | 8 weeks
  Dietary patterns and nutritional intake will be assessed at baseline and at Week 8. Participants will undergo an interview to assess compliance and tolerability at various time points (weeks 2, 5, and 8) throughout the 8-week feeding schedule.
Evaluate the effects of mixed beans on cognitive function | 16 weeks
  Data from the cognitive assessments collected at time 0 and Week 8 of the feeding schedule, and in follow-up post consumption at Weeks 2, 4, and 8, will be analyzed according to the statistical guide and recommendations provided with these tests. The cognitive tests that will be administered are: Mini Mental State Examination, Hopkins Verbal Learning, Digit Symbol Similarities Test, and Digit Span.

CONTACTS AND LOCATIONS:
Overall Officials: Peter C Zahradka, PhD, Principal Investigator — University of Manitoba
Locations (1):
- I.H Asper Clinical Research Institute, Winnipeg, Manitoba, Canada

REFERENCES:
- [Background] Dzau VJ, Braun-Dullaeus RC, Sedding DG. Vascular proliferation and atherosclerosis: new perspectives and therapeutic strategies. Nat Med. 2002 Nov;8(11):1249-56. doi: 10.1038/nm1102-1249. No abstract available. PMID 12411952
- [Background] Wilson PW, D'Agostino RB, Sullivan L, Parise H, Kannel WB. Overweight and obesity as determinants of cardiovascular risk: the Framingham experience. Arch Intern Med. 2002 Sep 9;162(16):1867-72. doi: 10.1001/archinte.162.16.1867. PMID 12196085
- [Background] Calkin AC, Allen TJ. Diabetes mellitus-associated atherosclerosis: mechanisms involved and potential for pharmacological invention. Am J Cardiovasc Drugs. 2006;6(1):15-40. doi: 10.2165/00129784-200606010-00003. PMID 16489846
- [Background] Juvenile Diabetes Research Foundation (2005) http://www jdrf org au/publications/factsheets/complications html
- [Background] Li TY, Rana JS, Manson JE, Willett WC, Stampfer MJ, Colditz GA, Rexrode KM, Hu FB. Obesity as compared with physical activity in predicting risk of coronary heart disease in women. Circulation. 2006 Jan 31;113(4):499-506. doi: 10.1161/CIRCULATIONAHA.105.574087. PMID 16449729
- [Background] British Heart Foundation Statistics (2006) www heartstats org
- [Background] Poels MM, van Oijen M, Mattace-Raso FU, Hofman A, Koudstaal PJ, Witteman JC, Breteler MM. Arterial stiffness, cognitive decline, and risk of dementia: the Rotterdam study. Stroke. 2007 Mar;38(3):888-92. doi: 10.1161/01.STR.0000257998.33768.87. Epub 2007 Feb 1. PMID 17272780
- [Background] Waldstein SR, Rice SC, Thayer JF, Najjar SS, Scuteri A, Zonderman AB. Pulse pressure and pulse wave velocity are related to cognitive decline in the Baltimore Longitudinal Study of Aging. Hypertension. 2008 Jan;51(1):99-104. doi: 10.1161/HYPERTENSIONAHA.107.093674. Epub 2007 Nov 19. PMID 18025297
- [Background] Houston DK, Stevens J, Cai J, Haines PS. Dairy, fruit, and vegetable intakes and functional limitations and disability in a biracial cohort: the Atherosclerosis Risk in Communities Study. Am J Clin Nutr. 2005 Feb;81(2):515-22. doi: 10.1093/ajcn.81.2.515. PMID 15699243
- [Background] Bazzano LA, Serdula MK, Liu S. Dietary intake of fruits and vegetables and risk of cardiovascular disease. Curr Atheroscler Rep. 2003 Nov;5(6):492-9. doi: 10.1007/s11883-003-0040-z. PMID 14525683
- [Background] Hu FB, Willett WC. Optimal diets for prevention of coronary heart disease. JAMA. 2002 Nov 27;288(20):2569-78. doi: 10.1001/jama.288.20.2569. PMID 12444864
- [Background] Anderson JW, Major AW. Pulses and lipaemia, short- and long-term effect: potential in the prevention of cardiovascular disease. Br J Nutr. 2002 Dec;88 Suppl 3:S263-71. doi: 10.1079/BJN2002716. PMID 12498626
- [Background] Castro IA, Barroso LP, Sinnecker P. Functional foods for coronary heart disease risk reduction: a meta-analysis using a multivariate approach. Am J Clin Nutr. 2005 Jul;82(1):32-40. doi: 10.1093/ajcn.82.1.32. PMID 16002797
- [Background] Rowland I. Optimal nutrition: fibre and phytochemicals. Proc Nutr Soc. 1999 May;58(2):415-9. doi: 10.1017/s0029665199000543. PMID 10466185
- [Background] Gylling H, Miettinen TA. The effect of plant stanol- and sterol-enriched foods on lipid metabolism, serum lipids and coronary heart disease. Ann Clin Biochem. 2005 Jul;42(Pt 4):254-63. doi: 10.1258/0004563054255605. PMID 15989725
- [Background] Hertog MG, Feskens EJ, Hollman PC, Katan MB, Kromhout D. Dietary antioxidant flavonoids and risk of coronary heart disease: the Zutphen Elderly Study. Lancet. 1993 Oct 23;342(8878):1007-11. doi: 10.1016/0140-6736(93)92876-u. PMID 8105262
- [Background] Keli SO, Hertog MG, Feskens EJ, Kromhout D. Dietary flavonoids, antioxidant vitamins, and incidence of stroke: the Zutphen study. Arch Intern Med. 1996 Mar 25;156(6):637-42. PMID 8629875
- [Background] Wylie-Rosett J, Segal-Isaacson CJ, Segal-Isaacson A. Carbohydrates and increases in obesity: does the type of carbohydrate make a difference? Obes Res. 2004 Nov;12 Suppl 2:124S-9S. doi: 10.1038/oby.2004.277. PMID 15601960
- [Background] Delzenne NM, Cani PD. A place for dietary fibre in the management of the metabolic syndrome. Curr Opin Clin Nutr Metab Care. 2005 Nov;8(6):636-40. doi: 10.1097/01.mco.0000171124.06408.71. PMID 16205465
- [Background] Matvienko OA, Lewis DS, Swanson M, Arndt B, Rainwater DL, Stewart J, Alekel DL. A single daily dose of soybean phytosterols in ground beef decreases serum total cholesterol and LDL cholesterol in young, mildly hypercholesterolemic men. Am J Clin Nutr. 2002 Jul;76(1):57-64. doi: 10.1093/ajcn/76.1.57. PMID 12081816
- [Background] Sharma RD. Isoflavones and hypercholesterolemia in rats. Lipids. 1979 Jun;14(6):535-9. doi: 10.1007/BF02533528. PMID 459719
- [Background] Cassidy A, Brown JE, Hawdon A, Faughnan MS, King LJ, Millward J, Zimmer-Nechemias L, Wolfe B, Setchell KD. Factors affecting the bioavailability of soy isoflavones in humans after ingestion of physiologically relevant levels from different soy foods. J Nutr. 2006 Jan;136(1):45-51. doi: 10.1093/jn/136.1.45. PMID 16365057
- [Background] Milerova J, Cerovska J, Zamrazil V, Bilek R, Lapcik O, Hampl R. Actual levels of soy phytoestrogens in children correlate with thyroid laboratory parameters. Clin Chem Lab Med. 2006;44(2):171-4. doi: 10.1515/CCLM.2006.031. PMID 16475902
- [Background] Huang Y, Cao S, Nagamani M, Anderson KE, Grady JJ, Lu LJ. Decreased circulating levels of tumor necrosis factor-alpha in postmenopausal women during consumption of soy-containing isoflavones. J Clin Endocrinol Metab. 2005 Jul;90(7):3956-62. doi: 10.1210/jc.2005-0161. Epub 2005 Apr 19. PMID 15840745
- [Background] Colacurci N, Chiantera A, Fornaro F, de Novellis V, Manzella D, Arciello A, Chiantera V, Improta L, Paolisso G. Effects of soy isoflavones on endothelial function in healthy postmenopausal women. Menopause. 2005 May-Jun;12(3):299-307. doi: 10.1097/01.gme.0000147017.23173.5b. PMID 15879919
- [Background] Heald CL, Bolton-Smith C, Ritchie MR, Morton MS, Alexander FE. Phyto-oestrogen intake in Scottish men: use of serum to validate a self-administered food-frequency questionnaire in older men. Eur J Clin Nutr. 2006 Jan;60(1):129-35. doi: 10.1038/sj.ejcn.1602277. PMID 16205743
- [Background] Ozasa K, Nakao M, Watanabe Y, Hayashi K, Miki T, Mikami K, Mori M, Sakauchi F, Washio M, Ito Y, Suzuki K, Kubo T, Wakai K, Tamakoshi A; JACC Study Group. Association of serum phytoestrogen concentration and dietary habits in a sample set of the JACC Study. J Epidemiol. 2005 Jun;15 Suppl 2(Suppl II):S196-202. doi: 10.2188/jea.15.s196. PMID 16127234
- [Background] Guillon F, Champ MM. Carbohydrate fractions of legumes: uses in human nutrition and potential for health. Br J Nutr. 2002 Dec;88 Suppl 3:S293-306. doi: 10.1079/BJN2002720. PMID 12498630
- [Background] Zahradka, P., Guzman, R., Weighell, W., Wright, B., Baldwin, A., Louis, S., Rodriguez, D., and Taylor, C.G. 2009 Increased consumption of legumes improves arterial stiffness in peripheral vascular disease independent of blood pressure, weight and serum cholesterol. Experimental Biology 2009, April 18-22, New Orleans, LA. [oral presentation].
- [Background] Pittaway JK, Ahuja KD, Chronopoulos A et al (2004) The effect of chickpeas on human serum lipids and lipoproteins. Asia Pac J Clin Nutr 13: S70
- [Background] He XZ, Reddy JT, Dixon RA. Stress responses in alfalfa (Medicago sativa L). XXII. cDNA cloning and characterization of an elicitor-inducible isoflavone 7-O-methyltransferase. Plant Mol Biol. 1998 Jan;36(1):43-54. doi: 10.1023/a:1005938121453. PMID 9484461
- [Background] Sumner LW, Paiva NL, Dixon RA, Geno PW. High-performance liquid chromatography/continuous-flow liquid secondary ion mass spectrometry of flavonoid glycosides in leguminous plant extracts. J Mass Spectrom. 1996 May;31(5):472-85. doi: 10.1002/(SICI)1096-9888(199605)31:53.0.CO;2-E. PMID 8799289
- [Background] Teede HJ, McGrath BP, DeSilva L, Cehun M, Fassoulakis A, Nestel PJ. Isoflavones reduce arterial stiffness: a placebo-controlled study in men and postmenopausal women. Arterioscler Thromb Vasc Biol. 2003 Jun 1;23(6):1066-71. doi: 10.1161/01.ATV.0000072967.97296.4A. Epub 2003 Apr 24. PMID 12714433
- [Background] DiCenzo GL, VanEtten HD. Studies on the late steps of (+) pisatin biosynthesis: evidence for (-) enantiomeric intermediates. Phytochemistry. 2006 Apr;67(7):675-83. doi: 10.1016/j.phytochem.2005.12.027. Epub 2006 Feb 28. PMID 16504226
- [Background] Tiemann K, Inze D, Van Montagu M, Barz W. Pterocarpan phytoalexin biosynthesis in elicitor-challenged chickpea (Cicer arietinum L.) cell cultures. Purification, characterization and cDNA cloning of NADPH:isoflavone oxidoreductase. Eur J Biochem. 1991 Sep 15;200(3):751-7. doi: 10.1111/j.1432-1033.1991.tb16241.x. PMID 1915347
- [Background] Robbins MP, Bolwell GP, Dixon RA. Metabolic changes in elicitor-treated bean cells. Selectivity of enzyme induction in relation to phytoalexin accumulation. Eur J Biochem. 1985 May 2;148(3):563-9. doi: 10.1111/j.1432-1033.1985.tb08877.x. PMID 3996394
- [Background] Ohkawara S, Okuma Y, Uehara T, Yamagishi T, Nomura Y. Astrapterocarpan isolated from Astragalus membranaceus inhibits proliferation of vascular smooth muscle cells. Eur J Pharmacol. 2005 Nov 21;525(1-3):41-7. doi: 10.1016/j.ejphar.2005.08.063. Epub 2005 Nov 16. PMID 16297381
- [Background] Rizkalla SW, Bellisle F, Slama G. Health benefits of low glycaemic index foods, such as pulses, in diabetic patients and healthy individuals. Br J Nutr. 2002 Dec;88 Suppl 3:S255-62. doi: 10.1079/BJN2002715. PMID 12498625
- [Background] Cazarolli LH, Zanatta L, Alberton EH, Figueiredo MS, Folador P, Damazio RG, Pizzolatti MG, Silva FR. Flavonoids: cellular and molecular mechanism of action in glucose homeostasis. Mini Rev Med Chem. 2008 Sep;8(10):1032-8. doi: 10.2174/138955708785740580. PMID 18782055
- [Background] Hooper L, Kroon PA, Rimm EB, Cohn JS, Harvey I, Le Cornu KA, Ryder JJ, Hall WL, Cassidy A. Flavonoids, flavonoid-rich foods, and cardiovascular risk: a meta-analysis of randomized controlled trials. Am J Clin Nutr. 2008 Jul;88(1):38-50. doi: 10.1093/ajcn/88.1.38. PMID 18614722
- [Background] American Heart Association Nutrition Committee; Lichtenstein AH, Appel LJ, Brands M, Carnethon M, Daniels S, Franch HA, Franklin B, Kris-Etherton P, Harris WS, Howard B, Karanja N, Lefevre M, Rudel L, Sacks F, Van Horn L, Winston M, Wylie-Rosett J. Diet and lifestyle recommendations revision 2006: a scientific statement from the American Heart Association Nutrition Committee. Circulation. 2006 Jul 4;114(1):82-96. doi: 10.1161/CIRCULATIONAHA.106.176158. Epub 2006 Jun 19. PMID 16785338
- [Derived] Wang L, Goldberg EM, Taylor CG, Zahradka P, Aliani M. Analyses of serum and urinary metabolites in individuals with peripheral artery disease (PAD) consuming a bean-rich diet: relationships with drug metabolites. Appl Physiol Nutr Metab. 2022 Mar;47(3):243-252. doi: 10.1139/apnm-2021-0495. Epub 2021 Oct 26. PMID 34699735
- See also: Website for Canadian Centre for Agri-food Research in Health and Medicine — http://www.ccarm.ca